CLINICAL TRIAL: NCT04963894
Title: Effects of Home Rehabilitation of Balance Based on Functional Exercises in People With Parkinson's Disease: Randomized Controlled Trial
Brief Title: Effects of Home Rehabilitation of Balance Based on Functional Exercises in People With Parkinson's Disease
Acronym: balanceHOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Valencia (Other)
Collaborators: Asociación Parkinson Valencia (Other)
Responsible Party: Principal Investigator, Constanza San Martín, Associate professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1686831
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Biomechanics of Balance; Biomechanics of gait; Functional rehabilitation; Functional assessment
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Subjects will participate in a baseline assessment session (T0) before rehabilitative treatment, followed by random allocation to the Experimental group (8 weeks of functional balance physiotherapy) or the Home control group (daily functional activity). After these 8 weeks, all the participants will develop a second assessment session (T1) and rested for the next 8 weeks to develop after that the follow-up assessment session (T2). At this time, patients from the Home control group will be switch to the Experimental group, and participants from the Experimental group will follow a 4-month of inactivity wash-out period. After this, they will carry out the T0, T1, and T2 evaluations following the Home control group protocol.
  Additionally, a third group of participants with Parkinson's disease who habitually developed conventional physiotherapy in a rehabilitation gym and in groups of 6 people, were evaluated (Conventional control group) at T0, T1 and T2.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home functional balance physiotherapy (Experimental): Participants perform physical therapy at home individually with a physical therapist. The experimental program of the study of balance exercise in functional context is implemented.
  Interventions: Other: Home functional balance physiotherapy
- Home functional daily activity (No Intervention): Participants stay in home without physiotherapy. Participants maintained their normal daily activities, which included housework, shopping, or daily walks.
- Conventional physiotherapy (Active Comparator): Participants perform physical therapy in a rehabilitation gym and in groups of 10 people. The conventional program of physiotherapy is implemented.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Home functional balance physiotherapy — Experimental physiotherapy program is carried out at home to improve the balance of people with Parkinson's disease through exercises that simulate everyday functional contexts.
  Arms: Home functional balance physiotherapy
Other: Conventional physiotherapy — Conventional control physiotherapy program is carried out face-to-face in a rehabilitation gym and in groups of 6 people. The conventional program of physiotherapy includes conventional therapeutic goals of rehabilitation in people with Parkinson's disease.
  Arms: Conventional physiotherapy

SUMMARY:
Balance rehabilitation programs in people with Parkinson's disease (PD) that include functional exercises, i.e. using tasks of daily living in training, show improvements in variables related to balance and gait. In previous studies, the advantage of taking into account the specificity of the task and the inclusion of specific objectives for the motor rehabilitation of people with PD has been observed. The interventions with the best results are usually carried out in hospital centers or rehabilitation gyms and, in groups of people.

Due to the situation experienced since last March 2020, due to the Covid-19 pandemic, group rehabilitation programs have been affected, especially in those pathologies that involve older age groups such as PD. For this reason, the need to transfer therapies to the home is considered, as well as to make people aware of the importance of continued rehabilitation, even from other settings. In the present study, we propose a rehabilitation program at home for people with Parkinson's disease based on balance with functional exercises, which will be compared with a home control group of people with PD that stay at home without any physical rehabilitation, and a conventional group physiotherapy program carried out in a rehabilitation gym in groups of 6 people. The effects of the experimental intervention and the control groups will be evaluated on outcomes related to balance using a dynamometric platform and outcomes related to gait through 3D photogrammetry.

DETAILED DESCRIPTION:
I. Objectives and Hypothesis

General objective: To determine if the effects of home rehabilitation of functional balance on the biomechanics of balance and gait, quality of life, cognitive status, and general physical performance are greater than the effects observed from the daily life activities at home, and from a conventional face-to-face group physiotherapy program.

Specific objectives:

1. To analyze the intra- and inter-rater reliability of the balance assessment in people with PD with dynamometric platforms performing functional tasks of daily life.
2. Determine the balance performance of people with PD in functional tasks before starting a physical therapy program.
3. Compare the immediate effects observed of the functional exercise-based rehabilitation program with the evaluated effects of a group rehabilitation program and with control participants staying at home without physical therapy.
4. Compare the observed medium-term effects (8-weeks) of the functional balance rehabilitation program with the observed medium-term effects of the conventional group physiotherapy program and with control participants who remain at home without a physiotherapy program.
5. Analyze the influence of the severity of the disease, using the Hoehn and Yahr scale and the Unified scale of Parkinson's disease, on the effects of the home rehabilitation program based on functional exercises.

II. General procedures

First, the approval of the Human Ethics Committee of the University of Valencia has been obtained. After managing the agreement with the Parkinson Valencia Association, the recruitment of participants will be carried out and, to those interested, an information sheet will be given with all the details of the study. Once the intention to participate has been confirmed, a first evaluation of the volunteers will be carried out to verify compliance with the proposed selection criteria. In this evaluation, the documents of informed consent and authorization for the use of images in scientific publications will be signed if required; In addition, at this time a code will be assigned to each participant to ensure their anonymity during the investigation to the evaluating staff and those in charge of randomization and data analysis.

People were recruited who, as a result of the COVID-19 pandemic had transferred home or telematically all their therapies related to Parkinson's disease, and on the other hand, were also recruited people who continued with therapies face-to-face. From the home volunteer participants, they will be divided by a sequence of random numbers provided by the IBM SPSS Statistics v.23 program into two groups: experimental group and home control group. Additionally, the volunteers who maintained their therapies outside the home made up the conventional control group.

The evaluator will not know the assignment of the participants. After randomization, it will be verified that the groups (experimental, home control, and conventional control group) do not differ significantly in their sociodemographic characteristics, and severity of the disease. The physiotherapist who will carry out the evaluations of the outcomes before and after the intervention period will be a different person from the professional who will evaluate the participation criteria. On the other hand, the intervention programs (experimental and conventional) will be carried out by two different physiotherapists. Both the assessment and the physiotherapy sessions do not contain invasive procedures and only require participants to perform therapeutic exercises adapted to the physical condition of people with PD.

The pre-intervention (T0), post-intervention (T1), and follow-up evaluations at 8 weeks (T2) will be carried out at the Faculty of Medicine of the University of Valencia, with the tools provided by the research group to which the main researcher of the project belongs. The interventions of the experimental group will take place at the home of each participant. The group control group sessions will be held at the Parkinson Valencia Association facilities.

III. Methodology

III.1. Study design

The proposed study consists of a single-blind, randomized clinical trial with crossover. The study protocol has been developed according to the SPIRIT 2013 statement.

Subjects will participate in a baseline assessment session (T0) before rehabilitative treatment, followed by random allocation to the Experimental group (8 weeks of functional balance physiotherapy) or the Home control group (daily functional activity). After these 8 weeks, all the participants will develop a second assessment session (T1) and rest for the next 8 weeks to later carry out the follow-up assessment session (T2). At this time, patients from the Home control group will be switch to the Experimental group, and participants from the Experimental group will follow a 4-month period of inactivity wash-out. After this, they will carry out the T0, T1, and T2 evaluations following the Home control group protocol.

Additionally, a third group of participants with Parkinson's disease who regularly receive conventional physiotherapy were evaluated (Conventional control group). The evaluation sessions will be before starting the usual rehabilitation program after the 2-months summer break (T0), after 8-weeks of rehabilitation (T1), and after 8-weeks of follow-up (T2). This group of participants will carry out the physiotherapy in the usual format, that is, in a rehabilitation gym and in groups of 6 people.

III.2 Participants

The initial recruitment should be 112 people.

Inclusion Criteria:

* To present diagnosis of idiopathic Parkinson's disease
* To have H&Y stage between I and IV
* To perform independent gait with or without technical assistance
* To have stable parkinsonian medication for at least 1 month prior to the start of the intervention.

Exclusion Criteria:

* To have other diseases that affect balance or walking
* To present other diagnosed neurological pathologies
* To present chronic uncontrolled diseases
* To participate in another physical rehabilitation program during the intervention period or 1 month before starting it
* To unknow one of the two official languages of the Valencian Community (Spain).

III.3 Assessment and outcomes

I. Outcomes collected from the biomechanical evaluation of the balance and movement of the pressure center:

1. Total displacement: distance to the origin of the platform from the center of pressures of the displacement vector described by the projection of the center of gravity (mm).
2. Angle of displacement: orientation of the displacement vector (º).
3. Dispersion of the center of pressures in the X and Y axes: dispersion of the displacement vector described by the projection of the center of gravity in the mediolateral and anteroposterior direction (mm).
4. Swept area: area in which the participant sway occurs, calculated from the start of the test to the end of it (mm2).
5. Average speed: average speed of the projection of the participant's center of gravity during the test, from the beginning to the end (m / s).
6. Mediolateral and anteroposterior displacement: maximum distance in mediolateral and anteroposterior directions during exercise (mm).
7. Maximum mediolateral and anteroposterior force: maximum force in anteroposterior and mediolateral directions exerted during exercise (N).
8. Maximum displacement (%): percentage with respect to the normality pattern (segmented by sex, age and height) of the displacement achieved in each of the directions when measuring the stability limits.
9. Reaction time: time taken by the participant to reach each of the stability limits (s).
10. Success: estimator of the participant's stability once the objective of each of the stability limits has been reached. It is calculated as a percentage of the points that fall within the objective with respect to the possible (%).
11. Skill: estimator of the adjustment in the follow-up carried out by the participant with his center of gravity on the moving target. It is represented as a percentage (%).

II. Outcomes collected from the biomechanical evaluation of gait:

1. Gait speed: distance traveled by the body per unit of time, in the direction considered. It is expressed in meters per second (m / s).
2. Stride length: distance measured between two consecutive supports of the same foot, heel support is the reference used. It is expressed in meters (m).
3. Stride duration: time elapsed while developing a full stride. It is expressed in seconds (s).
4. Cadence: number of steps performed in a time interval, its most commonly adopted unit being the step per minute (step / min).
5. Support time: time elapsed while the support phase is taking place. It is expressed as a percentage according to the time elapsed with respect to the gait cycle (%).
6. Oscillation time: time elapsed while the oscillation phase develops. It is expressed as a percentage according to the time elapsed with respect to the gait cycle (%).
7. Stride length: distance measured in the direction of progression, separating the initial landing of one foot from the initial landing of the contralateral foot. If the left stride length is defined, it would be defined as the distance measured between the heel contact of the right foot and the heel contact of the left foot. Expressed in meters (m).
8. Maximum dorsiflexion of the ankle joint in swing phase: maximum angle of ankle dorsiflexion reached during swing phase, expressed in degrees (°).
9. Maximum flexion of the knee joint in the swing phase: maximum angle of knee flexion reached during the swing phase, expressed in degrees (°).
10. Maximum extension of the hip joint in stance phase: maximum angle of hip extension reached during stance, expressed in degrees (°).
11. Maximum flexion of the hip joint in the swing phase: maximum angle of hip flexion reached during the swing phase, expressed in degrees (°).

III. Outcomes obtained from performing clinical scales and tests:

1. Unified Parkinson Disease Rating Scale motor (UPDRS-motor): score obtained from the motor section (III) of the UPDRS scale, which assesses the characteristic signs of the disease. Low scores indicate better motor function.
2. Mini Mental Parkinson test (MMP): score obtained on 32 points of the MMP cognitive screening. A high score corresponds to a better test result.
3. Frontal Assessment Battery (FAB): score achieved in the FAB executive functions assessment test. The maximum is 18 points; high scores represent better performance.
4. Scales for Outcomes in Parkinson's Disease-Cognition (SCOPA-COG): results obtained on 43 points of the SCOPA-COG scale on general cognitive functions. A higher score indicates a better cognitive level.
5. Mini-BESTest: score obtained with the abbreviated version of the BESTest out of 28 points. The higher the score, the better dynamic balance.
6. Tinetti Mobility Test (TMT): score obtained on the TMT balance and gait assessment scale. A high score reveals better performance in the test.
7. Parkinson's Disease Questionnaire (PDQ-39): score obtained on the PDQ-39 scale regarding the quality of life of people with PD. A lower score indicates a better perception of quality of life.
8. Hamilton Anxiety Rating Scale (HARS): score resulting from the HARS test; high scores indicate more severe anxiety.
9. Hamilton Depression Rating Scale (HDRS or HAM-D): score obtained from the HDRS scale.

III.4 Description of the interventions

1. Experimental intervention - Experimental group: consists of a specific home balance rehabilitation program for people with PD through functional tasks. The main strategy will be to break down a daily task into static and dynamic exercises, in order to experience an individualized progression within each physiotherapy session. Each session will last 1 hour and there will be two sessions a week for 8 weeks. In turn, the sessions will be divided into the warm-up phase (10 minutes), the central phase of functional balance training (45 minutes) and the final stretching phase (5 minutes). In the warm-up phase, other therapeutic objectives will be alternated to work during the sessions because the experimental program focuses on balance training.
2. Control interventions:

   * Conventional control group: they will carry out a conventional physiotherapy program which covers different objectives of the rehabilitation of people with PD (breathing exercises, dissociation of the waist, joint mobility, transfers and postural changes, strengthening exercises, and balance training and the March). Each session will last 1 hour and there will be two sessions a week for 8 weeks.The format of these sessions is in a group of 6 people in the Parkinson Valencia Association rehabilitation gym.
   * Home control group: the participants will stay at home doing the normal daily activities that include housework, shopping, and daily walks.

III.5 Sample size, randomization and blinding

To achieve the main objective proposed in this study, a total of 93 people diagnosed with PD will be recruited. This sample size has been determined using the G*Power v.3.1 to detect a difference between the groups (3), with a small-medium effect (f = 0.15), a statistical significance of 5% at the two-tailed level, and a power of 95%. If 20% of possible dropouts are also considered during the study, the initial recruitment should be 112 people.

An extern researcher who is not involved in the development of the study will perform the randomization process. Stratified randomization will be performed considering the Hoehn & Yahr stages and the cognitive state. Participants will be allocated accordingly to: 1) Experimental intervention or 2) Home control group. The treating physiotherapists thereafter be responsible for the management and organization of the appointments with participants. To ensure masking, the assessments and the treatments were performed by different therapists.

ELIGIBILITY:
Inclusion Criteria:

* To present diagnosis of idiopathic Parkinson's disease
* To have H&Y stage between I and IV
* To perform independent gait with or without technical assistance
* To have stable parkinsonian medication for at least 1 month prior to the start of the intervention.

Exclusion Criteria:

* To have other diseases that affect balance or walking
* To present other diagnosed neurological pathologies
* To present chronic uncontrolled diseases
* To participate in another physical rehabilitation program during the intervention period or 1 month before starting it
* To unknow one of the two official languages of the Valencian Community (Spain).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean swept area of the Centre of Pressure (COP) during the functional motor balance test (Romberg test with an arms task) | 4 months
  Area in which the participant sway occurs on the dynamometric platform, calculated by the movement of the COP from the start of the test to the end of it (mm2). During the motor functional test, the patient maintains balance while performing a task with the upper limbs below 90º of shoulder flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Constanza San Martín Valenzuela, PhD., Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - University of Valencia, Valencia
  - Asociación Parkinson Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The following results will be published in scientific journals:
  * Study protocol
  * Analysis of the reliability and repeatability of the evaluation
  * Results of the effects of the experimental rehabilitation program and its comparison with the effects achieved in the passive and active control groups.

REFERENCES:
- [Background] Stozek J, Rudzinska M, Pustulka-Piwnik U, Szczudlik A. The effect of the rehabilitation program on balance, gait, physical performance and trunk rotation in Parkinson's disease. Aging Clin Exp Res. 2016 Dec;28(6):1169-1177. doi: 10.1007/s40520-015-0506-1. Epub 2015 Dec 10. PMID 26661467
- [Background] Santos SM, da Silva RA, Terra MB, Almeida IA, de Melo LB, Ferraz HB. Balance versus resistance training on postural control in patients with Parkinson's disease: a randomized controlled trial. Eur J Phys Rehabil Med. 2017 Apr;53(2):173-183. doi: 10.23736/S1973-9087.16.04313-6. Epub 2016 Nov 23. PMID 27879959
- [Background] Atterbury EM, Welman KE. Balance training in individuals with Parkinson's disease: Therapist-supervised vs. home-based exercise programme. Gait Posture. 2017 Jun;55:138-144. doi: 10.1016/j.gaitpost.2017.04.006. Epub 2017 Apr 4. PMID 28445854
- [Background] Klamroth S, Steib S, Devan S, Pfeifer K. Effects of Exercise Therapy on Postural Instability in Parkinson Disease: A Meta-analysis. J Neurol Phys Ther. 2016 Jan;40(1):3-14. doi: 10.1097/NPT.0000000000000117. PMID 26655098
- [Background] Leavy B, Joseph C, Lofgren N, Johansson H, Hagstromer M, Franzen E. Outcome Evaluation of Highly Challenging Balance Training for People With Parkinson Disease: A Multicenter Effectiveness-Implementation Study. J Neurol Phys Ther. 2020 Jan;44(1):15-22. doi: 10.1097/NPT.0000000000000298. PMID 31834166
- [Background] Wallen MB, Hagstromer M, Conradsson D, Sorjonen K, Franzen E. Long-term effects of highly challenging balance training in Parkinson's disease-a randomized controlled trial. Clin Rehabil. 2018 Nov;32(11):1520-1529. doi: 10.1177/0269215518784338. Epub 2018 Jul 2. PMID 29962227
- [Background] Rennie L, Opheim A, Dietrichs E, Lofgren N, Franzen E. Highly challenging balance and gait training for individuals with Parkinson's disease improves pace, rhythm and variability domains of gait - A secondary analysis from a randomized controlled trial. Clin Rehabil. 2021 Feb;35(2):200-212. doi: 10.1177/0269215520956503. Epub 2020 Sep 28. PMID 32985265
- [Background] Liu C, Shiroy DM, Jones LY, Clark DO. Systematic review of functional training on muscle strength, physical functioning, and activities of daily living in older adults. Eur Rev Aging Phys Act. 1 de octubre de 2014;11(2):95-106.
- [Background] Serrao M, Pierelli F, Sinibaldi E, Chini G, Castiglia SF, Priori M, Gimma D, Sellitto G, Ranavolo A, Conte C, Bartolo M, Monari G. Progressive Modular Rebalancing System and Visual Cueing for Gait Rehabilitation in Parkinson's Disease: A Pilot, Randomized, Controlled Trial With Crossover. Front Neurol. 2019 Aug 29;10:902. doi: 10.3389/fneur.2019.00902. eCollection 2019. PMID 31543859